CLINICAL TRIAL: NCT00896831
Title: Therapeutic Efficacy of Oral L-Ornithine-L-Aspartate on Liver Cirrhosis and Minimal Encephalopathy: a Single Center Placebo Control Double Blind Study
Brief Title: Therapeutic Efficacy of Oral L-Ornithine-L-Aspartate on Minimal Encephalopathy
Acronym: PORTOALEGRE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Mário Reis Álvares-da-Silva, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08461
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Hepatic Encephalopathy
Keywords: minimal hepatic encephalopathy; L-ornithine-L-aspartate; psychometric test; critical flicker frequency; quality of life; Treatment; Health-related quality of life
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — ornithylaspartate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-ornithine-L-aspartate (Active Comparator): 5 g L-ornithine-L-aspartate (1 sachet) three times per day for 60 days
  Interventions: Drug: L-ornithine-L-aspartate
- placebo (Placebo Comparator): 5 g (1 sachet) of placebo comparator three times per day for 60 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-ornithine-L-aspartate — L-ornithine-L-aspartate: 5 g (1 sachet) three times per day for 60 days
  Arms: L-ornithine-L-aspartate
Drug: placebo — Placebo: 5 g (1 sachet) three times per day for 60 days
  Arms: placebo

SUMMARY:
The study aimed to assess the effectiveness and safety of L-ornithine-L-aspartate in the management of hepatic encephalopathy.

DETAILED DESCRIPTION:
Hepatic encephalopathy continues to be a major clinical problem in cirrhosis. Patients with minimal hepatic encephalopathy are at risk for accidents, had a decline in work performance, or complain of cognitive symptoms, with poor health-related quality of life. This study will compare L-ornithine-L-aspartate with placebo for 60 days to assess the effectiveness, safety and health-related quality of life of this drug.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis and diagnosis of minimal hepatic encephalopathy using psychometric tests and critical flicker frequency

Exclusion Criteria:

* Hepatic encephalopathy grade 1 to 4
* Use of drugs to treatment of hepatic encephalopathy (lactulose, neomycin)
* Psychoactive substance use within 72 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Psychometric tests and critical flicker frequency | day 0, 15, 30, 45 and 60

SECONDARY OUTCOMES:
Ammonia concentration | time 0 and 60 days after
Health-related quality of life | time 0 and 60 days after
Safety analysis | time 0 and 60 days after

CONTACTS AND LOCATIONS:
Overall Officials: Mário R Álvares-da-Silva, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil